CLINICAL TRIAL: NCT00944502
Title: Multicenter Clinical Study, Phase III, Prospective, Randomized, Double-blind, Comparative to Evaluate the Efficacy and Tolerability of the Use of Vitatonus Dexa Compared to Dexamethasone in Patients With Neuralgia of Various Origins
Brief Title: To Evaluate the Efficacy and Tolerability of the Use of Vitatonus Dexa Compared to Dexamethasone in Patients With Neuralgia of Various Origins
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bunker Industria Farmaceutica Ltda. (Industry)
Responsible Party: Elaine Pessoa, Bunker Indústria Farmacêutica Ltda.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E03-BUN-VITD-02/07
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Last update posted 2009-07-24 (Estimated); Status verified 2009-07

CONDITIONS: Neuralgia
Keywords: Neuralgy; Dexamethasone; Complex Vitamins; Injection; Symptoms of neuralgy of various origins
MeSH Terms: conditions — Neuralgia | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone and complex vitamins (Experimental): Group A: Vitatonus dexa injectable:
  1 ampoule intramuscularly every 3 days for 10 days.
  Group B: Vitatonus DEXA tablet:
  1 tablet orally every 8 hours for 10 days.
  Interventions: Drug: Dexamethasone
- Dexamethasone (Active Comparator): Group C: Dexamethasone Injectable:
  1 ampoule intramuscularly every 3 days for 10 days.
  Group D: Dexamethasone tablet:
  1 tablet orally every 8 hours for 10 days.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Group A: Vitatonus DEXA injectable:
  1 ampoule intramuscularly every 3 days for 10 days.
  Group B: Vitatonus DEXA tablets:
  1 tablet orally every 8 hours for 10 days.
  Group C: Dexamethasone Injectable:
  1 ampoule intramuscularly every 3 days for 10 days.
  Group D: Dexamethasone tablets:
  1 tablet orally every 8 hours for 10 days.
  Other Names: Vitatonus dexa tablest; Vitatonus Dexa Injectable

SUMMARY:
To evaluate the efficacy and tolerability of Vitatonus Dexa compared with dexamethasone in the signs and symptoms of neuralgia of various origins.

Clinical study, randomized prospective and random in nature, with a patients diagnosed with neuralgia of diverse origin.

Patients will be include in sufficient quantity to achieve the minimum of 104 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who consent to participate in the study by signing the ICF;
2. Patients of any ethnic group of both sexs aged over 18 years;
3. Patients with clinical diagnosis of neuralgia of various origins.
4. Patients who present scores on the Visual Analogue Scale (VAS) greater than or equal to 4 for PAIN.

Exclusion Criteria:

1. Patients with known hypersensitivity to lidocaine and thiamine or any component of the formula;
2. Pregnant women and nursing mothers;
3. Hypertensive or cardiac patients;
4. Patients with history of ulcers in the stomach or duodenum, diabetes mellitus or severe infections;
5. Patients who use levodopa, salicylates, colchicine, aminoglycosides, chloramphenicol, anticonvusivantes or potassium supplement.
6. Patient with a history of alcohol or use illicit drugs;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2009-10; Primary Completion 2009-11 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Observation of adverse events related to medication. The causality of adverse events concerning the use of medication will be given after applying the Naranjo Algorythm | Ten days

SECONDARY OUTCOMES:
Efficacy evaluation Likert scale and Visual Analogue | Ten days

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Hasan, Principal Investigator — Faculdade de Medicina do ABC
Locations (1):
- Faculdade de Medicina do ABC, Santo André, São Paulo, Brazil